CLINICAL TRIAL: NCT04756791
Title: Prospective Comparison of Single-Injection Serratus Anterior Plane Block With Ropivacaine Versus Local Infiltration of Anaesthetic After Breast Surgery
Acronym: SAPLIA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no participants recruited due to logistic problems
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAPLIA
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2023-05

CONDITIONS: Mastectomy; Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local infiltration anesthesia (Active Comparator): Patients will receive local infiltration anesthesia with ropivacaine placed by surgeon.
  Interventions: Procedure: Local Injection Anesthesia
- Serratus anterior plane block (Experimental): Patients receive a SAPB with ropivacaine placed by anesthesiologist.
  Interventions: Procedure: SAPB

INTERVENTIONS:
Procedure: SAPB — local anesthetic is injected between the serratus anterior and latissimus dorsi muscles.
  Arms: Serratus anterior plane block
Procedure: Local Injection Anesthesia — Anesthesia is injected directly into the tissue that is will be numbing.
  Arms: Local infiltration anesthesia

SUMMARY:
To evaluate whether a serratus anterior plane block (SAPB) is more effective than a local infiltration anesthesia (LIA) with an equal dose and same anesthetic performed by the surgeon, as an adjuvant to treat postoperative pain after unilateral mastectomy.

DETAILED DESCRIPTION:
To evaluate whether a serratus anterior plane block (SAPB) is more effective than a local infiltration anesthesia (LIA) with an equal dose and same anesthetic performed by the surgeon, as an adjuvant to treat postoperative pain after unilateral mastectomy.

Primary endpoint: the use of opioid's in the postoperative period. Secondary endpoint: Numerical Pain Rating Scale (NPRS) score recorded at the 2nd, 8th, 16th, 24th hour after surgery. 0 means no pain and 10 is the worst pain imaginable. In addition at the same time, we will look to the degree of arm mobilization where there will be 3 possible groups: 1. restricted, 2. fair mobilization and 3. free mobilization.

There are 2 treatment arms: 1st arm is the standard therapy, namely the local infiltration anesthesia. 2nd arm is the experimental arm, namely the SAPB. Patients are randomised into each arm after screening.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Provision of signed informed consent prior to any study-specific procedure.
* Patients who come to preoperative anesthesia consultation for their scheduled unilat-eral mastectomy.

Exclusion Criteria:

* Age >80 years
* History of chronic pain or drug treatment abuse
* Depression, psychiatric morbidity or mal-adaptive coping behavior
* Neuropathy
* Severe anxiety or other mental ailment, taking drugs affecting their capacity to assess pain
* Chronic or acute skin infection of the lateral thorax
* Hypersensitivity to ropivacaine
* Severe hepatic or renal disease
* Refuse to participate to the study
* Pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The use of opioids in the postoperative period | 24 hours
  Patients receive a patient controlled intravenous anesthesia pump with morphine. We will be able to analyze the total amount of opioid requested by the patient.

SECONDARY OUTCOMES:
Numerical Pain Rating Scale | 24 hours
  Patients will be asked at 4 different time points the amount of pain they are feeling on a scale of 0 to 10. 0 meaning no pain and 10 meaning the worst pain imaginable.
Degree of arm mobilization | 24 hours
  How much can the arm be mobilized of the patients? 3 groups: 1: restricted, 2: fair mobilization and 3. free mobilization

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided